#### Consent to Take Part in a Human Research Study

#### Title of research study:

# Innovation Labs for understanding and enhancing collaboration among early career scholars

**Version Date: 2018-03-06** 

#### Investigators:

Larry Hawk, Ph.D., Professor of Psychology, University at Buffalo

Timothy Murphy, M.D. SUNY Distinguished Professor of Medicine & Director, University at Buffalo Clinical and Translational Science Institute

#### Why am I being invited to take part in a research study?

You are being invited to take part in a research study because you are applying to participate in *Innovation Labs*.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, contact Dr. Hawk at <a href="mailto:lhawk@buffalo.edu">lhawk@buffalo.edu</a> or 716-645-0192. You may also contact the research participant advocate at 716-888-4845 or researchadvocate@buffalo.edu.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at (716) 888-4888 or email <u>ub-irb@buffalo.edu</u> if:

- You have questions about your rights as a participant in this research
- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team
- You want to talk to someone besides the research team.
- You want to get information or provide input about this research.

## Why is this research being done?

We aim to better understand attitudes and behavior related to collaboration among early career scholars and to evaluate the impact of week-long *Innovation Labs*.

## How long will the research last?

You will be in this research study for about 15 months. All applicants will be asked to complete electronic assessments at four time points, and each assessment will require about an hour. In addition, participants who attend the *Innovation Lab* will spend 5 full days at the *Lab* (~50 hours).

## How many people will be studied?

We expect between 100 and 200 applicants/participants, with approximately 25 selected to attend the *Innovation Lab*.

#### What happens if I say yes, I want to be in this research?

After providing your informed consent, you can submit your application. Once the application deadline closes, we will review complete applications for quality and diversity. From the resulting pool of highly qualified applicants, we will randomly select a subset to attend the *Innovation Lab*. All information you provide, including the application, will be used for research.

<u>Baseline assessment</u>. You will be asked to complete (within 2 weeks of the application deadline) a web-based survey about your scholarly activity and your attitudes towards collaboration and to submit your curriculum vitae and supplemental information about grant proposals, manuscripts and publications, and conference attendance and presentations. With the help of NCATS, your NIH eRA Commons ID may be used to gather additional information. You will be asked to provide information about social networking, and you will be provided with login credentials for an online community for early career scholars. You are not required to join, but if you do join, your activity on the site will be automatically captured as part of the project.

The baseline assessment is collected independently of the application. Although you must complete the baseline survey in order to be selected for the Innovation Lab, your specific responses to the survey will not be shared with the selection committee and will not influence the selection process in any way.

<u>Innovation Lab.</u> The <u>Innovation Lab</u> methodology was developed to counteract the myriad forces that push for monodisciplinary incremental science by fostering rapid but thoughtful development of innovative transdisciplinary research proposals. <u>Innovation Labs</u> follow the five stages of the creative problem-solving process: data gathering (Day 1), problem framing (Day 2), idea generation and "stretching" (Day 3), solution/proposal creation with real-time peer-review (Day 4), and action planning – development of detailed proposals (Day 5). Throughout the process, there is a deliberate focus on both expertise identification and the creation of strong social bonds between participants. Participants need not bring specific research ideas to the *Innovation Lab*. Rather, the ideas emerge through the application of the creative problem-solving process, in an organic and dynamic manner. A team of scientific experts or "mentors" play dual roles of coaches and reviewers, and facilitators guide the process.

If you are selected for the *Innovation Lab*, we will follow NIH guidelines in covering your lodging, airfare and per diem for the 5-day immersive workshop.

<u>Follow-up assessments</u>. All applicants will be asked to complete assessments similar to baseline assessment at approximately 3, 9, and 15 months after the baseline assessment.

# What happens if I do not want to be in this research?

Your participation in this research study is voluntary. You may choose not to enroll in this study. If you choose not to participate in the research study, you will not be eligible to participate in the Innovation Lab event.

### What happens if I say yes, but I change my mind later?

You can leave the research at any time, it will not be held against you.

## Is there any way being in this study could be bad for me?

Other than a potential confidentiality breach, which will be mitigated by using secure online data handling software (RedCap), there are no anticipated risks to participating in this research study.

#### Will being in this study help me in any way?

We cannot promise any benefits to you or others from your taking part in this research. However, participants in the *Innovation Lab* may establish new, productive collaborations as a result of this study. Information that is acquired and analyzed from this study will be made available to the public in aggregated form, and may contribute to the development of strong "best practices" for developing scientific collaborations among the translational workforce.

#### What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and education records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

For those who attend the Innovation Lab, a workshop designed to expand networks of connections, the fact of your attendance will not be confidential. This assures that participants and leaders in the Innovation Lab can introduce peers to each other, seek consultation, and connect via email, on social media, and through other platforms. It also allows us to share the names and affiliations of Innovation Lab attendees, as well as photos from the event, with other CTSAs, in our reports to the National Institutes of Health, and in promotional materials.

# Can I be removed from the research without my OK?

The principal investigator of the study can remove you from the research study without your approval. Possible reasons for removal include:

- We discover that a participant provided inaccurate information in the application process.
- A participant has not followed program requirements.
- The Sponsor, University, or Investigators have decided to stop the program.

#### What else do I need to know?

If you participate, we will compensate for completing the follow-up assessments: \$50 each for the 3-, 9-, and 15-month follow-ups. If you complete all three follow-up assessments within 2 weeks of our requests, you will receive a \$50 bonus along with the compensation for the 15-month follow-up. If you are selected for the *Innovation Lab*, we will follow NIH guidelines and pay for your lodging and meals during the workshop and reimburse you for airfare and ground transportation. covering your lodging, airfare and per diem for the 5-day immersive workshop. (Complete details and instructions are available on the application website.)

This study is sponsored by the National Center for the Advancement of Translational Research.

| By entering your initials and the date below<br>will be indicating your consent to participat | |
|---|---|
| Initials: Today's date: | o ar anno rocomion projecti |